CLINICAL TRIAL: NCT01816776
Title: A Randomized Trial Evaluating the Safety and Effectiveness of the remedē® System in Patients With Central Sleep Apnea
Brief Title: Respicardia, Inc. Pivotal Trial of the remedē System
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Respicardia, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Respicardia CR-1005
Record Dates: First submitted 2013-03-19; First posted 2013-03-22 (Estimated); Results first posted 2017-07-11 (Actual); Last update posted 2018-06-29 (Actual); Status verified 2018-05

CONDITIONS: Sleep Apnea, Central; Sleep Disordered Breathing; Heart Failure
MeSH Terms: conditions — Sleep Apnea, Central; Sleep Apnea Syndromes; Heart Failure | interventions — Control Groups

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Treatment Group (Experimental): Subjects implanted with the remedē system device and randomized to the Treatment group will receive optimal medical therapy and have the remedē system initiated to deliver transvenous stimulation of the phrenic nerve at the Therapy Initiation Visit (1 month post device implant).
  Interventions: Device: Treatment Group (transvenous stimulation of the phrenic nerve)
- Control group (Other): Subjects implanted with the remedē system device and randomized to the Control group will receive optimal medical therapy through the 6-month Post-Therapy Initiation Visit. Control group subjects will have the remedē system initiated to deliver transvenous stimulation of the phrenic nerve at the 6-month Post-Therapy Initiation Visit (7 months post device implant).
  Interventions: Device: Control Group (Optimal Medical Therapy)

INTERVENTIONS:
Device: Treatment Group (transvenous stimulation of the phrenic nerve) — device implant, optimal medical therapy and device initiation 1 month post implant.
  Other Names: remedē System; Transvenous stimulation of the phrenic nerve
  Arms: Treatment Group
Device: Control Group (Optimal Medical Therapy) — device implant, optimal medical therapy and delayed device initiation (7 months post device implant)
  Other Names: Optimal Medical Therapy
  Arms: Control group

SUMMARY:
The primary purpose of this prospective, multicenter, randomized trial is to evaluate the safety and effectiveness of therapy delivered by the remedē® system in subjects with moderate to severe central sleep apnea and optimal medical management, compared to outcomes in randomized control subjects receiving optimal medical management and implanted but inactive remedē® systems.

ELIGIBILITY:
Inclusion Criteria:

1. At least 18 years of age
2. Central Sleep apnea confirmed by core lab analysis of PSG with EEG within 40 days of scheduled implant:

   * Apnea/Hypopnea Index (AHI) greater than or equal to 20;
   * Central Apnea Index (CAI) at least 50% of all apneas, with at least 30 central apnea events;
   * Oxygen Desaturation Index (OAI) less than or equal to 20% of the total AHI
3. Medically stable for 30 days prior to all baseline testing (including PSG), i.e., no hospitalizations for illness, no breathing mask-based therapy, and on stable medications and therapies:

   * Stable medications are defined as no changes during this period except for those within a pre-specified sliding scale medication regimen;
   * If the subject has heart failure, the baseline testing (including PSG) should occur at least 6 months after initial diagnosis;
   * If the subject has systolic heart failure, the baseline testing (including PSG) should occur after maximally titrating beta blockers, angiotensin converting enzyme inhibitors (ACE-I) and other medications indicated in the current guidelines (unless contraindicated or not considered medically necessary) and after receiving any indicated device therapy including devices for cardiac resynchronization therapy and/or primary prevention of sudden cardiac death;
   * If subject has a hospitalization or physician visit requiring IV medication between the screening PSG and implant, the subject must be re-screened when stable
4. Expected to tolerate study procedures in the opinion of the investigator, in particular:

   * Ability to lie down long enough to insert the remede system without shortness of breath and able to tolerate instrumentation for the Polysomnogram/Polygram testing;
   * Expected to tolerate therapy titration and the sensation of therapy, and communicate therapy experience.
5. In the investigator's opinion, willing and able to comply with all study requirements
6. Signed the Institutional Review Board/Medical Ethics Committee approved informed consent (HIPAA authorization in the U.S.)

Exclusion Criteria:

1. Pacemaker dependent subjects without any physiologic escape rhythm
2. Suspected inability to place catheter for delivery of stimulation lead (e.g. previously know coagulopathy, distorted anatomy, prior failed pectoral implant, etc.)
3. Evidence of phrenic nerve palsy
4. More than 2 previous open chest surgical procedures (e.g., CABG)
5. Etiology of central sleep apnea known to be caused primarily by pain medication
6. Documented history of psychosis or severe bipolar disorder
7. Cerebrovascular accident (CVA) within 12 months of baseline testing
8. History of idiopathic pulmonary hypertension, World Health Organization Class 1
9. Limited pulmonary function with either forced expiratory volume (FEV) 1/forced vital capacity (FVC) less than 65% of predicted value or FVC less than 60% of predicted value
10. Baseline oxygen saturation less than 92% while awake and on room air after 5 minutes of quiet rest
11. Anticipated need for chronic oxygen therapy or breathing mask-based therapy for 6 months post therapy initiation visit
12. Active infection or sepsis within 30 days of enrollment
13. Currently on renal dialysis or creatinine level greater than 2.5 mg/dL or calculated creatinine clearance equal to or less than 30 ml/min using the Cockcroft-Gault equation
14. Poor liver function with baseline aspartate transaminase (AST), alanine transaminase (ALT), and/or total bilirubin greater than 3 times the upper limit of normal (per lab normals at each site)
15. Hemoglobin less than 8 gm/dL
16. In subjects with heart failure, American College of Cardiology (ACC)/American Heart Association Heart (AHA) Stage D
17. Within the 3 months prior to baseline testing, any of the following: uncorrected severe valvular stenosis, valve replacement or repair (percutaneous or surgical), myocardial infarction (MI), coronary artery bypass grafting (CABG) surgery, percutaneous coronary intervention (PCI), cardiac ablation, new cardiac resynchronization device or new pacemaker implant
18. New implantable cardioverter defibrillator or any implantable device generator change-out within 30 days prior to baseline testing or anticipated within the first 6 months of enrollment
19. Other anticipated surgery or invasive procedure expected to affect ability to perform testing at 6-month post-therapy initiation visit
20. Unstable angina
21. Allergy to or intolerant of contrast dye
22. Pregnancy or of child bearing potential without a negative pregnancy test within 10 days prior to remede system implant
23. Life expectancy or expected time to transplant or left ventricular assist device of less than 12 months
24. Currently enrolled or planning to enroll in another study that may conflict with protocol requirements or confound subject results in this trial

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 151 (Actual)
Dates: Start 2013-03; Primary Completion 2016-09-10 (Actual); Study Completion 2017-11-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Maria Rosa Costanzo, M.D., Principal Investigator — Midwest Heart Specialists
Locations (30):
- United States (23):
  - Keck Hospital of USC, Los Angeles, California
  - University of Florida - Jacksonville, Jacksonville, Florida
  - Advocate Medical Group, Downers Grove, Illinois
  - Edward Hospital-Advocate Medical Group, Naperville, Illinois
  - University of Maryland, Baltimore, Baltimore, Maryland
  - Johns Hopkins Bayview Medical Center, Baltimore, Maryland
  - Detroit Clinical Research Center, Farmington Hills, Michigan
  - Spectrum Health, Grand Rapids, Michigan
  - United Heart and Vascular (Allina), Saint Paul, Minnesota
  - Mid America Heart Institute, Kansas City, Missouri
  - Washington University, St Louis, Missouri
  - Bryan Heart, Lincoln, Nebraska
  - Cooper Health System, Cherry Hill, New Jersey
  - Novant Medical Group, Inc. Presbyterian Sleep Health Charlotte, Charlotte, North Carolina
  - Forsyth Medical Center - Novant, Winston-Salem, North Carolina
  - The Lindner Center for Research and Education at Christ Hospital, Cincinnati, Ohio
  - Ohio State University, Columbus, Ohio
  - Lancaster General Hospital, Lancaster, Pennsylvania
  - Hospital of University of Pennsylvania, Philadelphia, Pennsylvania
  - Stern Cardiovascular, Memphis, Tennessee
  - Methodist Healthcare System, San Antonio, Texas
  - Virginia Commonwealth University, Richmond, Virginia
  - Marshfield Clinic, Marshfield, Wisconsin
- Germany (6):
  - Bad Oeynhausen- Heart & Diabetes Center, Bad Oeynhausen
  - Charite Medical School, Campus Virchow-Klinikum, Berlin
  - Bernau-Herzzentruym Brandenburg, Bernau
  - Bielefeld-Klinikun, Bielefeld
  - Hamburg: Universitares Herzzentrum, Hamburg
  - Ambulantes Herzzentrum-Kassel, Kassel
- Fourth Military Hospital, Wroclaw, Poland

REFERENCES:
- [Derived] Javaheri S, McKane SW, Germany RE. Changes in quality of life in patients with atrial fibrillation and central sleep apnea treated with transvenous phrenic nerve stimulation. Sleep Med. 2026 Feb 2;141:108824. doi: 10.1016/j.sleep.2026.108824. Online ahead of print. PMID 41643229
- [Derived] Dupuy-McCauley K, Schwartz AR, Javaheri S, Germany R, McKane S, Morgenthaler TI. Classifying hypopneas as obstructive or central can enhance transvenous phrenic nerve stimulation therapy patient selection and outcomes. J Clin Sleep Med. 2025 Dec 1;21(12):2113-2120. doi: 10.5664/jcsm.11904. PMID 41025409
- [Derived] Samii S, McKane S, Meyer TE, Shah N. Analysis by sex of safety and effectiveness of transvenous phrenic nerve stimulation. Sleep Breath. 2024 Mar;28(1):165-171. doi: 10.1007/s11325-023-02882-5. Epub 2023 Jul 12. PMID 37436669
- [Derived] Baumert M, Linz D, McKane S, Immanuel S. Transvenous phrenic nerve stimulation is associated with normalization of nocturnal heart rate perturbations in patients with central sleep apnea. Sleep. 2023 Sep 8;46(9):zsad166. doi: 10.1093/sleep/zsad166. PMID 37284759
- [Derived] Costanzo MR, Javaheri S, Ponikowski P, Oldenburg O, Augostini R, Goldberg LR, Stellbrink C, Fox H, Schwartz AR, Gupta S, McKane S, Meyer TE, Abraham WT; remede(R)System Pivotal Trial Study Group. Transvenous Phrenic Nerve Stimulation for Treatment of Central Sleep Apnea: Five-Year Safety and Efficacy Outcomes. Nat Sci Sleep. 2021 Apr 29;13:515-526. doi: 10.2147/NSS.S300713. eCollection 2021. PMID 33953626
- [Derived] Schwartz AR, Goldberg LR, McKane S, Morgenthaler TI. Transvenous phrenic nerve stimulation improves central sleep apnea, sleep quality, and quality of life regardless of prior positive airway pressure treatment. Sleep Breath. 2021 Dec;25(4):2053-2063. doi: 10.1007/s11325-021-02335-x. Epub 2021 Mar 20. PMID 33745107
- [Derived] Javaheri S, McKane S. Transvenous phrenic nerve stimulation to treat idiopathic central sleep apnea. J Clin Sleep Med. 2020 Dec 15;16(12):2099-2107. doi: 10.5664/jcsm.8802. PMID 32946372
- [Derived] Costanzo MR. Central Sleep Apnea in Patients with Heart Failure-How to Screen, How to Treat. Curr Heart Fail Rep. 2020 Oct;17(5):277-287. doi: 10.1007/s11897-020-00472-0. PMID 32803641
- [Derived] Oldenburg O, Costanzo MR, Germany R, McKane S, Meyer TE, Fox H. Improving Nocturnal Hypoxemic Burden with Transvenous Phrenic Nerve Stimulation for the Treatment of Central Sleep Apnea. J Cardiovasc Transl Res. 2021 Apr;14(2):377-385. doi: 10.1007/s12265-020-10061-0. Epub 2020 Aug 12. PMID 32789619
- [Derived] Fox H, Oldenburg O, Javaheri S, Ponikowski P, Augostini R, Goldberg LR, Stellbrink C, Mckane S, Meyer TE, Abraham WT, Costanzo MR. Long-term efficacy and safety of phrenic nerve stimulation for the treatment of central sleep apnea. Sleep. 2019 Oct 21;42(11):zsz158. doi: 10.1093/sleep/zsz158. PMID 31634407
- [Derived] Costanzo MR, Ponikowski P, Javaheri S, Augostini R, Goldberg L, Holcomb R, Kao A, Khayat RN, Oldenburg O, Stellbrink C, Abraham WT; remede System Pivotal Trial Study Group. Transvenous neurostimulation for central sleep apnoea: a randomised controlled trial. Lancet. 2016 Sep 3;388(10048):974-82. doi: 10.1016/S0140-6736(16)30961-8. Epub 2016 Sep 1. PMID 27598679
- [Derived] Costanzo MR, Augostini R, Goldberg LR, Ponikowski P, Stellbrink C, Javaheri S. Design of the remede System Pivotal Trial: A Prospective, Randomized Study in the Use of Respiratory Rhythm Management to Treat Central Sleep Apnea. J Card Fail. 2015 Nov;21(11):892-902. doi: 10.1016/j.cardfail.2015.08.344. PMID 26432647

RESULTS

PARTICIPANT FLOW:
Groups:
- Treatment Group: Subjects implanted with the remedē System device who receive optimal medical therapy and remedē System therapy.
- Control Group: Subjects implanted with the remedē System device who receive optimal medical therapy alone (remedē System inactive through 6 months).
Period: Overall Study
Arm/Group | Treatment Group | Control Group
Started (Randomized) | 73 | 78
6 Month Primary Effectiveness Assessed | 68 | 73
Completed (Primary safety assessed through 12 months) | 60 | 70
Not Completed | 13 | 8

BASELINE CHARACTERISTICS:
Population: Intent-to-treat
Groups:
- Total: Total of all reporting groups
Arm/Group | Treatment Group | Control Group | Total
Number analyzed (Participants) | 73 | 78 | 151
Age, Continuous [Mean (Standard Deviation); unit: years] | 65 (12) | 65 (13) | 65 (13)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10 | 6 | 16
  Male | 63 | 72 | 135
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 4 | 5
  Not Hispanic or Latino | 72 | 74 | 146
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 3 | 3 | 6
  White | 70 | 74 | 144
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 1 | 1
Region of Enrollment [Number; unit: participants]
  United States | 49 | 50 | 99
  Poland | 10 | 11 | 21
  Germany | 14 | 17 | 31
Apnea-Hypopnea Index (AHI) [Mean (Standard Deviation); unit: Events/hour] — The number of apneas and hypopneas per hour of sleep.
  An apnea is defined by 3 characteristics:
  1. There is a drop in the peak thermal sensor excursion or alternate nasal air pressure transducer (inspiratory effort) by > 90% of baseline
  2. The duration of the event lasts at least 10 seconds
  3. At least 90% of the event's duration meets the amplitude reduction criteria for apnea
  Hypopnea defined as 30% reduction in airflow (or alternative hypopnea sensor) for ≥10 seconds over at least 90% of the event's duration that is associated with a >4% fall in oxygen saturation from baseline.
  Events/hour | 48.8 (19.3) | 43.7 (16.8) | 46.2 (18.2)
Central Apnea Index (CAI) [Mean (Standard Deviation); unit: Events/hour] — The number of central apneas per hour of sleep. A central apnea is defined by 4 characteristics:
  1. There is a drop in the peak thermal sensor excursion or alternate nasal air pressure transducer (inspiratory effort) by > 90% of baseline
  2. The duration of the event lasts at least 10 seconds
  3. At least 90% of the event's duration meets the amplitude reduction criteria for apnea
  4. An apnea associated with absent inspiratory effort throughout the period
  Events/hour | 30.0 (18.0) | 26.6 (16.1) | 28.2 (17.1)
Arousal Index (ArI) [Mean (Standard Deviation); unit: Events/hour] — The number of arousals per hour of sleep. During sleep stages N1, N2, N3 or rapid eye movement (REM), an abrupt shift of electroencephalogram frequency including alpha, theta and/or frequencies greater than 16 Hz that last at least 3 seconds, with at least 10 seconds of stable sleep preceding the change is an arousal.
  Events/hour | 45.5 (17.9) | 43.6 (19.1) | 44.6 (18.5)
Rapid Eye Movement Sleep (REM) [Mean (Standard Deviation); unit: Percent] — REM is a sleep stage. The percentage of sleep in REM is a measure of sleep quality.
  Percent | 10.4 (7.2) | 11.8 (7.1) | 11.1 (7.1)
Oxygen Desaturation Index (ODI4) [Mean (Standard Deviation); unit: Events/hour] — Number of times per hour of sleep that the blood's oxygen level drops by ≥4%.
  Events/hour | 43.2 (21.7) | 37.5 (17.5) | 40.2 (19.8)
Obstructive Apnea Index [Mean (Standard Deviation); unit: Events/hour] — The number of obstructive apneas per hour of sleep. An obstructive apnea is defined by 4 characteristics:
  1. There is a drop in the peak thermal sensor excursion or alternate nasal air pressure transducer (inspiratory effort) by > 90% of baseline
  2. The duration of the event lasts at least 10 seconds
  3. At least 90% of the event's duration meets the amplitude reduction criteria for apnea
  4. An apnea associated with continued or increased inspiratory effort throughout the period
  Events/hour | 2.6 (3.2) | 2.3 (2.7) | 2.4 (3.0)
Epworth Sleepiness Scale (ESS) [Mean (Standard Deviation); unit: units on a scale] — The ESS is an assessment to measure a subject's general level of daytime sleepiness. Scores can range from 0-24, with higher scores indicating higher level of daytime sleepiness.
  units on a scale | 10.2 (5.2) | 9.5 (5.8) | 9.8 (5.5)
Body mass index (BMI) [Mean (Standard Deviation); unit: kg/m2] | 30.8 (5.3) | 31.3 (6.6) | 31.1 (6.0)
Hypertension [Count of Participants; unit: Participants] | 53 | 60 | 113
Heart failure [Count of Participants; unit: Participants] — Defined as New York Heart Association (NYHA) Functional Class ≥ I
  Participants | 48 | 48 | 96
Left ventricular ejection fraction [Mean (Standard Deviation); unit: Percent] — Available for N=71 Treatment and N=75 Control participants. Population: Ejection fraction data not available on all subjects
  Percent
    number analyzed (Participants) | 71 | 75 | 146
    (all) | 39.7 (12.1) | 39.4 (12.2) | 39.6 (12.1)
Atrial fibrillation [Count of Participants; unit: Participants] | 32 | 32 | 64
Stroke [Count of Participants; unit: Participants] | 6 | 6 | 12
Coronary artery disease [Count of Participants; unit: Participants] | 40 | 44 | 84
Concomitant implantable device delivering therapy [Count of Participants; unit: Participants] | 31 | 33 | 64

OUTCOME MEASURES:

1. Primary Outcome: The Proportion of Participants Experiencing a Reduction in Apnea-hypopnea Index (AHI)
Description: Comparison of the proportion of subjects in the Treatment group achieving a 50% or greater reduction in AHI from baseline to 6 months compared to the Control group.
Time Frame: 6 months
Population: The population analyzed included all randomized participants who had a 6 month assessment. In addition, Treatment group subjects who did not have a 6 month assessment for reasons related to implant, device or delivered therapy were included as not achieving the endpoint.
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment Group | Control Group
Number analyzed (Participants) | 68 | 73
Participants | 35 | 8
Statistical Analysis 1: Comparison: Treatment Group vs Control Group; Test type: Superiority; p < 0.0001, Fisher Exact — 1-sided. p<0.025 considered significant; Risk Difference (RD) = 41, 95% CI 2-sided [25 to 54] — Risk difference = Treatment - Control

2. Primary Outcome: Freedom From Related Serious Adverse Events Within 12 Months
Description: Freedom from serious adverse events (SAEs) associated with the implant procedure, the remede System, or the delivered therapy at 12 months post therapy initiation visit.
Time Frame: 12 months
Population: Intent-to-treat. The study protocol pre-specified that randomized groups be combined to assess freedom from related serious adverse events within 12 months.
Measure: Count of Participants; unit: Participants
Groups:
- Pooled Group: All randomized participants pooled. All subjects were implanted with the remedē System device and received optimal medical therapy. The Treatment group had received 12 months active therapy and Control had received 6 months active therapy.
Arm/Group | Pooled Group
Number analyzed (Participants) | 151
Participants | 138

3. Secondary Outcome: Central Apnea Index (CAI) Change From Baseline at 6 Months
Description: Change in CAI = Month 6 index - Baseline index. The central apnea index is a measurement used to indicate the severity of central sleep apnea. It is represented by the number of central apnea events per hour of sleep.
Time Frame: 6 months
Population: Per protocol: excludes patients who did not meet major entry criteria, had therapy programmed to "off" at the 6-month visit, did not have 6-month polysomnogram (PSG) results or had unsuccessful implant attempt.
Measure: Mean (95% Confidence Interval); unit: Events/hour
Arm/Group | Treatment Group | Control Group
Number analyzed (Participants) | 58 | 73
Events/hour | -25.7 [-30.5 to -21.0] | -2.9 [-7.0 to 1.2]
Statistical Analysis 1: Comparison: Treatment Group vs Control Group; Test type: Superiority; p < 0.0001, Wilcoxon (Mann-Whitney) — 1-sided. Secondary endpoints hierarchically tested with p<0.025 considered significant; Mean Difference (Net) = -22.8, 95% CI 2-sided [-29.0 to -16.6] — Mean difference = Treatment - Control

4. Secondary Outcome: Apnea-Hypopnea Index (AHI) Change From Baseline at 6 Months
Description: Change in AHI = Month 6 index - Baseline index. The Apnea-Hypopnea Index is a measurement used to indicate the severity of sleep apnea. It is represented by the number of apnea and hypopnea events per hour of sleep.
Time Frame: 6 months
Population: Per protocol: excludes patients who did not meet major entry criteria, had therapy programmed to "off" at the 6-month visit, did not have 6-month PSG results or had unsuccessful implant attempt.
Measure: Mean (95% Confidence Interval); unit: Events/hour
Arm/Group | Treatment Group | Control Group
Number analyzed (Participants) | 58 | 73
Events/hour | -23.9 [-28.8 to -19.0] | 1.1 [-3.0 to 5.2]
Statistical Analysis 1: Comparison: Treatment Group vs Control Group; Test type: Superiority; p < 0.0001, t-test, 1 sided — Secondary endpoints hierarchically tested with p<0.025 considered significant; Mean Difference (Net) = -25.0, 95% CI 2-sided [-31.2 to -18.7] — Mean difference = Treatment - Control

5. Secondary Outcome: Arousal Index (ArI) Change From Baseline at 6 Months
Description: Change in ArI = Month 6 index - Baseline index. The Arousal Index is a measurement used to indicate the number of times per hour of sleep that sleep is disrupted.
Time Frame: 6 months
Population: as for outcome 4
Measure: Mean (95% Confidence Interval); unit: Events/hour
Arm/Group | Treatment Group | Control Group
Number analyzed (Participants) | 58 | 73
Events/hour | -20.2 [-25.2 to -15.2] | -5.0 [-9.2 to -0.8]
Statistical Analysis 1: Comparison: Treatment Group vs Control Group; Test type: Superiority; p < 0.0001, t-test, 1 sided — Secondary endpoints hierarchically tested with p<0.025 considered significant; Mean Difference (Net) = -15.2, 95% CI 2-sided [-21.6 to -8.7] — Mean difference = Treatment - Control

6. Secondary Outcome: Rapid Eye Movement (REM) Sleep Change From Baseline at 6 Months
Description: Change in REM = Month 6 percentage - Baseline percentage. Rapid Eye Movement (REM) is a sleep stage. A higher percentage of sleep in REM is a measure of better sleep quality.
Time Frame: 6 months
Population: as for outcome 4
Measure: Mean (95% Confidence Interval); unit: percentage of sleep
Arm/Group | Treatment Group | Control Group
Number analyzed (Participants) | 58 | 73
percentage of sleep | 1.8 [-0.3 to 4.0] | -0.6 [-2.4 to 1.3]
Statistical Analysis 1: Comparison: Treatment Group vs Control Group; Test type: Superiority; p = 0.0244, Wilcoxon (Mann-Whitney) — 1-sided. Secondary endpoints hierarchically tested with p<0.025 considered significant; Mean Difference (Net) = 2.4, 95% CI 2-sided [-0.4 to 5.1] — Mean difference = Treatment - Control

7. Secondary Outcome: The Proportion of Participants Experiencing a Marked or Moderate Improvement in Patient Global Assessment at 6 Months
Description: The proportion of subjects with a "moderate" or "marked" improvement in the Patient Global Assessment from baseline to the 6 month visit
Time Frame: 6 months
Population: Per protocol: excludes patients who did not meet major entry criteria, had therapy programmed to "off" at the 6-month visit, did not have 6-month PSG results or had unsuccessful implant attempt. Note: 1 Control subject did not provide a response and is excluded from analysis.
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment Group | Control Group
Number analyzed (Participants) | 58 | 72
Participants | 35 | 4
Statistical Analysis 1: Comparison: Treatment Group vs Control Group; Test type: Superiority; p < 0.0001, Fisher Exact — 1-sided. Secondary endpoints hierarchically tested with p<0.025 considered significant; Risk Difference (RD) = 55, 95% CI 2-sided [40 to 68] — Risk difference = Treatment - Control

8. Secondary Outcome: Oxygen Desaturation Index 4% (ODI4) Change From Baseline at 6 Months
Description: Change in ODI4 = Month 6 index - Baseline index. The Oxygen Desaturation Index 4% is a measurement of the number of times per hour of sleep that the blood's oxygen level drops ≥4%.
Time Frame: 6 months
Population: as for outcome 4
Measure: Mean (95% Confidence Interval); unit: Events/hour
Arm/Group | Treatment Group | Control Group
Number analyzed (Participants) | 58 | 73
Events/hour | -19.1 [-23.9 to -14.3] | 3.6 [-0.5 to 7.6]
Statistical Analysis 1: Comparison: Treatment Group vs Control Group; Test type: Superiority; p < 0.0001, t-test, 1 sided — Secondary endpoints hierarchically tested with p<0.025 considered significant; Mean Difference (Net) = -22.7, 95% CI 2-sided [-28.9 to -16.5] — Mean difference = Treatment - Control

9. Secondary Outcome: Epworth Sleepiness Scale (ESS) Change From Baseline at 6 Months
Description: Change in ESS = Month 6 score - Baseline score. The ESS is an assessment to measure a subject's general level of daytime sleepiness. Scores can range from 0-24, with higher scores indicating higher level of daytime sleepiness.
Time Frame: 6 months
Population: as for outcome 4
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Treatment Group | Control Group
Number analyzed (Participants) | 58 | 73
units on a scale | -3.6 [-5.1 to -2.1] | 0.1 [-0.9 to 1.2]
Statistical Analysis 1: Comparison: Treatment Group vs Control Group; Test type: Superiority; p < 0.0001, Wilcoxon (Mann-Whitney) — 1-sided. Secondary endpoints hierarchically tested with p<0.025 considered significant; Mean Difference (Net) = -3.7, 95% CI 2-sided [-5.5 to -2.0] — Mean difference = Treatment - Control

ADVERSE EVENTS:
Time Frame: Implant through 12 Months post therapy initiation visit window
Groups:
- Pooled Group: The study protocol pre-specified that randomized groups be combined to assess safety. All subjects were implanted with the remedē System device and received optimal medical therapy. The Treatment group had received 12 months active therapy and Control had received 6 months active therapy.
Arm/Group | Pooled Group
All-Cause Mortality (participants affected / at risk) | 7/151
Serious Adverse Events (participants affected / at risk) | 74/151
Other Adverse Events (participants affected / at risk) | 53/151
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Pooled Group (N=151)
ANEMIA (Blood and lymphatic system disorders) | 2
HEART FAILURE (Cardiac disorders) | 16
SUSTAINED VENTRICULAR TACHY ARRHYTHMIA (Cardiac disorders) | 11
ATRIAL FIBRILLATION (Cardiac disorders) | 5
AORTIC VALVE DISEASE (Cardiac disorders) | 3
CORONARY ARTERY DISEASE (Cardiac disorders) | 3
CHEST PAIN - CARDIAC (Cardiac disorders) | 2
COMPLICATION OF HEART FAILURE THERAPY (Cardiac disorders) | 2
MYOCARDIAL INFARCTION (Cardiac disorders) | 2
ACUTE CORONARY SYNDROME (Cardiac disorders) | 1
ATRIAL FLUTTER (Cardiac disorders) | 1
COMPLICATION OF CARDIAC SURGERY (Cardiac disorders) | 1
INAPPROPRIATE ICD SHOCK (Cardiac disorders) | 1
MITRAL VALVE DISEASE (Cardiac disorders) | 1
PERICARDIAL EFFUSION (Cardiac disorders) | 1
RIGHT HEART PERFORATION (Cardiac disorders) | 1
SICK SINUS SYNDROME (Cardiac disorders) | 1
SUDDEN DEATH (Cardiac disorders) | 1
DIABETIC KETOACIDOSIS (Endocrine disorders) | 1
DIABETIC TOE (Endocrine disorders) | 1
GASTROESOPHAGEAL REFLUX DISEASE (Gastrointestinal disorders) | 2
COLONIC PERFORATION (Gastrointestinal disorders) | 1
DIVERTICULITIS (Gastrointestinal disorders) | 1
GASTROINTESTINAL BLEED SECONDARY TO WARFARIN (Gastrointestinal disorders) | 1
GASTROPARESIS (Gastrointestinal disorders) | 1
INGUINAL HERNIA (Gastrointestinal disorders) | 1
PERFORATED BOWEL (Gastrointestinal disorders) | 1
IMPENDING POCKET EROSION (General disorders) | 3
IMPLANT SITE INFECTION (General disorders) | 2
NON-CARDIAC CHEST PAIN (General disorders) | 2
STIMULATION LEAD DISLODGEMENT (REMEDE SYSTEM) (General disorders) | 2 — The stimulation lead pulled out of the target vessel and required the lead to be replaced in order to deliver therapy
ABDOMINAL DISCOMFORT (General disorders) | 1
ALTERED MENTAL STATUS (General disorders) | 1
CONCOMITANT DEVICE INTERACTION (General disorders) | 1
DEGENERATIVE JOINT DISEASE (General disorders) | 1
ELECTIVE EXPLANT OF REMEDE SYSTEM (General disorders) | 1
EXTRA-RESPIRATORY STIMULATION (General disorders) | 1 — Discomfort of feeling delivered therapy in areas remote from the diaphragm
FLU LIKE SYMPTOMS (General disorders) | 1
ICD LEAD FAILURE (General disorders) | 1
IMPLANT SITE HEMATOMA (General disorders) | 1
SINUS INFECTION (General disorders) | 1
STIMULATION LEAD COMPONENT FAILURE (REMEDE SYSTEM) (General disorders) | 1
STIMULATION LEAD DISPLACEMENT (REMEDE SYSTEM) (General disorders) | 1 — The stimulation lead remained in the target vessel but electrode position did not allow for effective therapy delivery
SEPSIS (Infections and infestations) | 3
PNEUMONIA (Infections and infestations) | 2
BLADDER INFECTION (Infections and infestations) | 1
BRONCHIAL INFECTION (Infections and infestations) | 1
CELLULITIS (Infections and infestations) | 1
DIABETIC FOOT INFECTION (Infections and infestations) | 1
ENDOCARDITIS INFECTIVE (Infections and infestations) | 1
ICD IMPLANT SITE INFECTION (Infections and infestations) | 1
LEG CELLULITIS (Infections and infestations) | 1
FRACTURE (Injury, poisoning and procedural complications) | 3
AORTIC INJURY (Injury, poisoning and procedural complications) | 1
INTRAOPERATIVE NEUROLOGICAL INJURY (Injury, poisoning and procedural complications) | 1
ELEVATED TRANSAMINASE (Investigations) | 1
DEHYDRATION (Metabolism and nutrition disorders) | 1
HYPERGLYCEMIA (Metabolism and nutrition disorders) | 1
HYPOGLYCEMIA (Metabolism and nutrition disorders) | 1
ARTHRITIS (Musculoskeletal and connective tissue disorders) | 2
BACK PAIN (Musculoskeletal and connective tissue disorders) | 2
BICEP TENDON TEAR (Musculoskeletal and connective tissue disorders) | 1
MENISCUS TEAR (Musculoskeletal and connective tissue disorders) | 1
RHABDOMYOLOSIS (Musculoskeletal and connective tissue disorders) | 1
ADENOCARCINOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
LUNG CANCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
MYELODYSPLASTIC SYNDROME (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
PROSTATE CARCINOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
STROKE (Nervous system disorders) | 2
AMNESIA (Nervous system disorders) | 1
ENCEPHALOPATHY (Nervous system disorders) | 1
HEADACHE (Nervous system disorders) | 1
MEMORY IMPAIRMENT (Nervous system disorders) | 1
SEIZURE (Nervous system disorders) | 1
TRANSIENT ISCHEMIC ATTACKS (Nervous system disorders) | 1
ACUTE KIDNEY INJURY (Renal and urinary disorders) | 1
URINARY TRACT STENOSIS (Renal and urinary disorders) | 1
DYSPNEA (Respiratory, thoracic and mediastinal disorders) | 1
PULMONARY EDEMA (Respiratory, thoracic and mediastinal disorders) | 1
RESPIRATORY FAILURE (Respiratory, thoracic and mediastinal disorders) | 1
CRT-D IMPLANT (Surgical and medical procedures) | 1
CYCLOPHOTOCOAGULATION (Surgical and medical procedures) | 1
DRUG ELUTING STENT (Surgical and medical procedures) | 1
ICD GENERATOR AND RV LEAD REPLACEMENT (Surgical and medical procedures) | 1
ICD IMPLANT (Surgical and medical procedures) | 1
LEFT SUBTALAR JOINT ARTHRODESIS, HARDWARE REMOVAL AND BONE GRAFTING (Surgical and medical procedures) | 1
TOOTH EXTRACTION (Surgical and medical procedures) | 1
HYPOTENSION (Vascular disorders) | 2
PULMONARY EMBOLISM (Vascular disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Pooled Group (N=151)
DIAPHRAGMATIC STIMULATION DISCOMFORT (General disorders) | 38 — Discomfort in the abdominal area due to remede System delivered therapy
EXTRA-RESPIRATORY STIMULATION (General disorders) | 14 — Discomfort of feeling delivered therapy in areas remote from the diaphragm
PAIN IN EXTREMITY (Musculoskeletal and connective tissue disorders) | 11

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No